CLINICAL TRIAL: NCT06698380
Title: The Effect of Mirror Therapy on Upper Extremity Motor Function in Stroke Rehabilitation
Acronym: MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Karthick Balasubramanian, Lecturer, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUREC-Apr.13/COM-2022/32-5
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Chronic Stroke Patients; Hemiplegia
Keywords: storke; Hemiplegia; mirror therapy; upper extremity; motor function
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The participants of control participants received conventional Physical Therapy (CPT) based on their routine physical therapy neurological evaluation. The CPT was individualized based on the needs of the subjects. It included: normalization of muscle tone, strengthening of weak muscles, lengthening of tight muscles, training for transfers like supine to sit, sit to stand, balance training, and gait training. The upper extremity training for ADLs also were incorporated using mobilization, reaching, grasping and dexterity movements
  Interventions: Other: Conventional Physical Therapy
- Experimental (Experimental): The experimental group received combination therapy that is MT combined with CPT treatment. The subjects were asked to be seated on a comfortable chair with feet and back supported and the upper extremity was on a tabletop surface of two-by-two- meter size.
  A mirror was positioned in front of the subjects to shield the involved upper extremity, reflecting the image of the uninvolved side. The involved upper extremity was placed in a relaxed posture beside the mirror, mirroring the same posture on the uninvolved side to enhance illusional movements. The MT for the experimental group included reaching, grasping, and dexterity movements of the unaffected upper limb, followed by imitation on the involved side. Subjects performed five activities: finger flexion and extension, finger opposition, counting with fingers, wrist flexion and extension, and forearm supination and pronation. Each activity was done 10 times, with mirror therapy lasting 15 minutes and 30 minutes / 6 weeks.
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Conventional Physical Therapy — The subjects of the control group received the CPT based on their routine physical therapy neurological evaluation. The CPT was individualized based on the needs of the subjects. It included: normalization of muscle tone, strengthening of weak muscles, lengthening of tight muscles, training for transfers like supine to sit, sit to stand, balance training, and gait training. The upper extremity training for ADLs also were incorporated using mobilization, reaching, grasping and dexterity movements
  Arms: Control
Other: Mirror Therapy — A mirror was positioned in front of the subjects to shield the involved upper extremity, reflecting the image of the uninvolved side. The involved upper extremity was placed in a relaxed posture beside the mirror, mirroring the same posture on the uninvolved side to enhance illusional movements. The MT for the experimental group included reaching, grasping, and dexterity movements of the unaffected upper limb, followed by imitation on the involved side. Subjects performed five activities: finger flexion and extension, finger opposition, counting with fingers, wrist flexion and extension, and forearm supination and pronation. Each activity was done 10 times, with mirror therapy lasting 15 minutes followed by 30 minutes of CPT treatment. Each session lasted 45 minutes, held three times per week over six weeks.
  Arms: Experimental

SUMMARY:
The study aimed to determine the effect of mirror therapy versus conventional physical therapy treatment in improving upper extremity impairments and motor function among chronic hemiplegic subjects.

Research Objectives:

1. To discover the effectiveness of conventional physical therapy treatment on improving upper limb motor function among chronic hemiplegic subjects.
2. To find out the effect of mirror therapy along with conventional physical therapy treatment on improving upper limb motor function among chronic hemiplegic subjects.
3. To find out the effectiveness of mirror therapy combined with conventional physical therapy treatment versus conventional physical therapy treatment alone on improving upper extremity motor function among chronic hemiplegic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Duration of stroke more than six months
* Subjects of chronic stroke with left or right hemiplegia.
* Genders of male and female with age ranging between forty-five to sixty-five years.
* MMSE scores greater than 23 out of 30.
* Scored one or one plus on MAS on all muscles of the affected upper limb.
* Have normal visual perception.
* Able to follow oral commands.

Exclusion Criteria:

* Unable to follow visual and oral commands.
* Unilateral neglect.
* Cognitive impairments (MMSE scores less than 24 out of 30), or language deficits.
* Any other neurological disorders and recent surgeries.
* Previous exposure to MT.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity (FMA-UE) | week 0 and week 6
  The most widely applied method in post-stroke rehabilitation to estimate gross motor impairment is the FMA. It pursues the concept of stages of recovery for stroke patients, which developed with Twitchell and Brunnstrom. It gauges the capacity to manage isolated joints, which are impeded by synergy, and the strength of muscle, with an assumed order of difficulty. The components of the assessment are five including: joint range of motion (ROM), balance, sensory function, motion of the joint, and joint discomfort. FMA-UE is split into whole, proximal, and distal components and these subtests investigate the movement of body parts independently, with the authors recommending that every part of UE heal alone. It is used in the clinical field and in research to detect disease progress, prescribe exercise recovery, and prepare and evaluate medicine. FMA has as well demonstrated excellent inter- and intra-rater reliability, also the feasibility of construction.
Wolf Motor Function Test (WMFT) | week 0 and week 6
  This examination tool was designed to estimate and evaluate the exercise capacity of individuals who suffer from mild to acute upper extremity motion impairments in laboratory and clinical settings. It is an improvement of a previous examination tool utilized in high-functioning patients, but difficult to perform in patients with minimal capacity of movement in the hands and fingers. WMFT has proven its significance in describing motion status in terms of severity and upper extremity motion impairments in a cohort of chronic individuals who suffer from stroke and traumatic brain injury in high-functioning individuals. The inter-test and inter-rater reliability, internal consistency of tests, and stability for schedule measures of performance and functional ability were high, varying from 0.88 to 0.98, with most estimates' relative from 0.95

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided